CLINICAL TRIAL: NCT00786305
Title: Assessment of Efficiency of Nebulized Ceftazidime and Amikacin in Treatment of Ventilator Associated Pneumonia Caused by Pseudomonas Aeruginosa
Brief Title: Nebulized Ceftazidime and Amikacin in Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Jean-Jacques Rouby, Groupe Hospitalier Pitie-Salpetriere
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NATB-2004
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Pneumonia
Keywords: Nebulization; ceftazidime; amikacin; pneumonia; Pseudomonas aeruginosa; mechanical ventilation; Ventilator-associated pneumonia; treatment
MeSH Terms: conditions — Pneumonia; Pseudomonas Infections; Pneumonia, Ventilator-Associated | interventions — Ceftazidime; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: nebulized ceftazidime and amikacin (Experimental)
  Interventions: Drug: ceftazidime and amikacin
- 2: intravenous ceftazidime and amikacin (Active Comparator)
  Interventions: Drug: ceftazidime and amikacin

INTERVENTIONS:
Drug: ceftazidime and amikacin — Nebulized ceftazidime 15 mg/kg/3h during 8 days and nebulized amikacin 25 mg/kg/day during 3 days
  Other Names: fortum and amiklin
  Arms: 1: nebulized ceftazidime and amikacin
Drug: ceftazidime and amikacin — Intravenous infusion of ceftazidime 30 mg/kg over 30 min followed by continuous infusion 90 mg/kg/day during 8 days and intravenous infusion of amikacin 15 mg/kg/day over 30 min during 3 days
  Other Names: fortum and amiklin
  Arms: 2: intravenous ceftazidime and amikacin

SUMMARY:
Pseudomonas aeruginosa is one of the major causative microorganisms of ventilator-associated pneumonia often resistant to antibiotics. In experimental models, nebulization of antibiotics delivers high lung tissue concentrations of antibiotics in infected lungs and increases lung bacterial killing. The aim of the study is to assess the efficiency of nebulized ceftazidime and amikacin in the treatment of pneumonia caused by Pseudomonas aeruginosa in ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years old, ventilator associated pneumonia caused by pseudomonas aeruginosa
* Written informed consent provided by the relatives

Exclusion Criteria:

* Pseudomonas aeruginosa resistant to ceftazidime and amikacin
* Pseudomonas aeruginosa pneumonia associated with other infections requiring intravenous treatment
* Severe septic shock and severe hypoxemia
* Allergy to ceftazidime or amikacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-10; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Bacterial killing | 14 days

SECONDARY OUTCOMES:
Changes of lung aeration | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Rouby, MD, PhD, Principal Investigator — La Pitie-Salpetriere hospital
Locations (1):
- Intensive care unit, Department of anesthesiology, La pitie-Salpetriere hospital, Paris, France